CLINICAL TRIAL: NCT07228052
Title: Giving Asthmatics Intramuscular Steroids for Preventing Return to the Emergency Department: A Randomized Control Trial
Brief Title: Giving Asthmatics Intramuscular Steroids for Preventing Return to the Emergency Department
Acronym: GASPING
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-16648
Record Dates: First submitted 2025-11-12; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: dexamethasone; prednisone; randomized controlled trial
MeSH Terms: conditions — Asthma | interventions — Dexamethasone; Prednisone

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned 1:1 to a treatment group using a computer-generated randomization schedule.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, treating physicians, nursing, and the investigators will remain blinded to treatment allocation. Blinded medications will be pre-packaged by the clinical research pharmacy team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Intramuscular Steroid Injection (Active Comparator): Dexamethasone 16mg Intramuscular Single Dose
  Interventions: Drug: Dexamethasone 16mg IM
- Oral Steroid Short Course (Active Comparator): Prednisone 60mg PO for 5 Days
  Interventions: Drug: Prednisone 60mg PO

INTERVENTIONS:
Drug: Dexamethasone 16mg IM — Dexamethasone 16mg Intramuscular Administration Once
  Arms: Single Intramuscular Steroid Injection
Drug: Prednisone 60mg PO — Prednisone 60mg PO for 5 Days
  Arms: Oral Steroid Short Course

SUMMARY:
This study aims to compare the efficacy of a one-time IM dose of dexamethasone versus a 5-day course of prednisone in adult ED patients presenting with asthma exacerbations. This is a randomized, controlled, double-blind, non-inferiority trial conducted at two urban EDs within the Montefiore Health System.

DETAILED DESCRIPTION:
Asthma exacerbations are a leading cause of emergency department (ED) visits in the United States. In pediatric patients, a single dose of dexamethasone has been widely adopted as an effective and convenient alternative to multi-day oral steroid regimens. However, in adults, evidence regarding the efficacy of a single-dose steroid approach compared to a traditional 5-day course of oral prednisone is mixed. Despite the availability of oral corticosteroids like prednisone, medication adherence after ED discharge remains a significant challenge. Studies indicate that only about 30% of ED patients fill prescribed medications post-discharge. A single-dose intramuscular (IM) dexamethasone regimen offers the advantage of ensuring adequate anti-inflammatory effects for asthma exacerbations. This study aims to compare the efficacy of a one-time IM dose of dexamethasone versus a 5-day course of prednisone in adult ED patients presenting with asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old presenting to the ED with an asthma exacerbation
* Diagnosed with asthma per International Classification of Diseases, 10th Revision (ICD-10) criteria or by the treating clinician
* Discharged from the ED with a primary diagnosis of asthma exacerbation
* Initiated systemic corticosteroids during the ED visit
* Must be English or Spanish speaking

Exclusion Criteria:

* Current use of systemic corticosteroids, including Emergency Medical Services (EMS) administration before ED arrival
* History of severe adverse reactions to corticosteroids
* Heart failure and uncontrolled diabetes (glucose >300mg/dL in the ED)
* Pregnancy or breastfeeding as prednisone is the preferred treatment for asthma in this population
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test Score | Within 4 Weeks post-discharge, up to 28-30 days
  Asthma control will be assessed via administration of the Asthma Control Test (ACT) questionnaire at 4 weeks post-discharge. The ACT questionnaire is comprised of 5 questions which ask participants to recall how asthma symptoms have affected them over the prior 4 weeks. Responses to the 5 questions are rated on a 5-point Likert scale ranging from 1-5, yielding an overall possible scoring range of 5-25. Higher ACT scores are indicative of better asthma control. For this study, an ACT score >19 indicates well-controlled asthma. Scores will be summarized by study arm using basic descriptive statistics.

SECONDARY OUTCOMES:
ED or Hospitalization for Asthma | Within 4 Weeks post-discharge, up to 28-30 days
  The number of return visits to the ED or hospitalizations related to asthma, within 30 days post-discharge, will be summarized by study arm using basic descriptive statistics.
Change in Quality of Life | At 2 weeks (at approximately 14-15 days) and 4 weeks post-discharge relative to baseline, up to 28-30 days
  Change in Quality of Life will be measured using the Mini Asthma Quality of Life Questionnaire (MiniAQLQ). The MiniAQLQ is a 21-item survey which consists of questions spanning four domains: symptoms, activity limitations, emotional function, and environmental stimuli, in order to understand how asthma affects patients in daily life. Responses to the first 15 questions are rated on a 7-point scale ranging from 1-7, questions 16-20 are rated using a 3-point scale ranging from 1-3, and question 21 is rated on 0-10 scale, with higher scores being indicative of a better quality of life, yielding an overall possible scoring range of 20-130. Scores will be summarized by study arm.
Adverse Effects | At Day 0 and 4-weeks post-discharge relative to baseline, up to 28-30 days
  Documented occurrence of Adverse Effects, including nausea, headache, rash, or Serious Adverse Events, as defined by International Conference on Harmonisation - Good Clinical Practice (ICH GCP) guidelines, will be summarized by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lutz, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Hasegawa K, Craig SS, Teach SJ, Camargo CA Jr. Management of Asthma Exacerbations in the Emergency Department. J Allergy Clin Immunol Pract. 2021 Jul;9(7):2599-2610. doi: 10.1016/j.jaip.2020.12.037. Epub 2020 Dec 31. PMID 33387672
- [Background] Keeney GE, Gray MP, Morrison AK, Levas MN, Kessler EA, Hill GD, Gorelick MH, Jackson JL. Dexamethasone for acute asthma exacerbations in children: a meta-analysis. Pediatrics. 2014 Mar;133(3):493-9. doi: 10.1542/peds.2013-2273. Epub 2014 Feb 10. PMID 24515516
- [Background] Kirkland SW, Cross E, Campbell S, Villa-Roel C, Rowe BH. Intramuscular versus oral corticosteroids to reduce relapses following discharge from the emergency department for acute asthma. Cochrane Database Syst Rev. 2018 Jun 2;6(6):CD012629. doi: 10.1002/14651858.CD012629.pub2. PMID 29859017
- [Background] Fischer MA, Jones JB, Wright E, Van Loan RP, Xie J, Gallagher L, Wurst AM, Shrank WH. A randomized telephone intervention trial to reduce primary medication nonadherence. J Manag Care Spec Pharm. 2015 Feb;21(2):124-31. doi: 10.18553/jmcp.2015.21.2.124. PMID 25615001
- [Background] Gordon S, Tompkins T, Dayan PS. Randomized trial of single-dose intramuscular dexamethasone compared with prednisolone for children with acute asthma. Pediatr Emerg Care. 2007 Aug;23(8):521-7. doi: 10.1097/PEC.0b013e318128f821. PMID 17726409
- [Background] Qureshi F, Zaritsky A, Poirier MP. Comparative efficacy of oral dexamethasone versus oral prednisone in acute pediatric asthma. J Pediatr. 2001 Jul;139(1):20-6. doi: 10.1067/mpd.2001.115021. PMID 11445789
- [Background] Nelsen LM, Kosinski M, Rizio AA, Jacques L, Schatz M, Stanford RH, Svedsater H. A structured review evaluating content validity of the Asthma Control Test, and its consistency with U.S. guidelines and patient expectations for asthma control. J Asthma. 2022 Mar;59(3):628-637. doi: 10.1080/02770903.2020.1861624. Epub 2020 Dec 30. PMID 33377411
- [Background] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Background] Alzahrani YA, Becker EA. Asthma Control Assessment Tools. Respir Care. 2016 Jan;61(1):106-16. doi: 10.4187/respcare.04341. Epub 2015 Nov 10. PMID 26556901
- [Background] Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009 Oct;124(4):719-23.e1. doi: 10.1016/j.jaci.2009.06.053. Epub 2009 Sep 19. PMID 19767070